CLINICAL TRIAL: NCT05581381
Title: Exploring the Effect of Empathy Training Program for Nurses
Brief Title: Empathy Training Program for Nursing Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Xuan-Yi Huang, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20210106R
Record Dates: First submitted 2022-10-07; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Empathy
Keywords: Nurses; Empathy Training Program; Effectiveness; Subjective Experience

STUDY DESIGN:
Intervention Model Description: The quantitative method is the experimental research method using randomization. The nurses receiving the intervention of empathy training program are in the experimental group, while those who do not receive it are in the control group. The effectiveness assessment will use the Empathy Construct Rating Scale (ECRS) and learning satisfaction scale, Empathy Construct Rating Scale (ECRS) required to be completed by both the experimental group and control group. ECRS perform the pre-test and post-test assessments. The pre-test perform before the implementation of empathy training program, and perform the post-test at week 8 the end of empathy training program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional empathy training program (Experimental): Provide empathy training for the experimental group for a total of 8 weeks (1 time a week, 1 hour each time).In the 8th week, both the experimental group and the control group must fill in the ECRS Empathy Scale; the experimental group must fill in the Learning Satisfaction Scale
  Interventions: Behavioral: empathy training program
- No intervention empathy training program (No Intervention): The control group did not offer empathy training.In the 8th week, both the experimental group and the control group must fill in the ECRS Empathy Scale.

INTERVENTIONS:
Behavioral: empathy training program — Empathy training, a total of 8 weeks of training (1 time a week, 1 hour each time)
  Arms: Interventional empathy training program

SUMMARY:
The research purpose is to investigate the effectiveness of empathy training program for nurses, as well as to investigate the effectiveness of learning satisfaction for nurses and the empathy training program learning subjective experience of nurses.The quantitative method is the experimental research method using randomization. The nurses receiving the intervention of empathy training program are in the experimental group, while those who do not receive it are in the control group.

DETAILED DESCRIPTION:
"Empathy" is an important foundation for nurses to communicate with patients and establish trust relationships. If nurses lack of empathy literacy or cannot apply empathy communication skills, the role of establishing therapeutic interpersonal relationships with patients or family members will affect the professional performance of nurses and the quality of nursing care. Therefore, improving nurses' empathy literacy and practical application ability has a great correlation with good care quality. However, domestic and international research on the correlation of empathy for nurses are not enough and lack of training program, which show the topic of this research is worth exploring.

The research purpose is to investigate the effectiveness of empathy training program for nurses, as well as to investigate the effectiveness of learning satisfaction for nurses and the empathy training program learning subjective experience of nurses.

In order to make the evaluation of research effectiveness more specific and objective, and also hoped that nurses can be the subject of effectiveness evaluation, and have a deeper understanding of their subjective experiences and feelings. Therefore, the effectiveness evaluation of empathy training program for nurses is using method triangulation of the qualitative and quantitative research method.

The quantitative method is the experimental research method using randomization. The nurses receiving the intervention of empathy training program are in the experimental group, while those who do not receive it are in the control group. The effectiveness assessment will use the Empathy Construct Rating Scale (ECRS) and learning satisfaction scale, Empathy Construct Rating Scale (ECRS) required to be completed by both the experimental group and control group. ECRS perform the pre-test, post-test and post-post-test assessments. The pre-test perform before the implementation of empathy training program, and perform the post-test at week 8 the end of empathy training program, and after 8 weeks of post-test performed the post-post-test. Only experimental group require to complete learning satisfaction scale, perform the post-test at week 8 the end of empathy training program. Descriptive phenomenological research method is used as the qualitative method to explore the empathy training program learning subjective experience of nurses. This study will use purposive sampling to enroll experimental group who has received empathy training program learning, and then perform individual in-depth interviews after the end of empathy training program. Non-structured interview guides are used.

Hopefully, this study may develop an empathy training program which is suitable for nurses. This can enhance the empathy literacy and practical application ability for nurses.

ELIGIBILITY:
Inclusion Criteria:

1. Nursing staff

Exclusion Criteria:

1. Nursing staff on night shifts
2. Nursing staff working in the hospice and psychiatric wards

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Empathy Construct Rating Scale | Pre-test
  A total of 56 questions . It has good reliability and validity (the internal consistency is 0.92, and the test reliability after two weeks is 0.95). The ECRS(Empathy Construct Rating Scale) includes four subscales of caring (38-item), empathy (9-item), professional relationship (5-item), and communication (4-item), which are scored on a Likert scale ranging from 1 (completely unsatisfactory) to 6 (full compliance), Higher scores indicate higher empathy
Empathy Construct Rating Scale | Post-test at Week 8
  A total of 56 questions . It has good reliability and validity (the internal consistency is 0.92, and the test reliability after two weeks is 0.95). The ECRS(Empathy Construct Rating Scale) includes four subscales of caring (38-item), empathy (9-item), professional relationship (5-item), and communication (4-item), which are scored on a Likert scale ranging from 1 (completely unsatisfactory) to 6 (full compliance), Higher scores indicate higher empathy

SECONDARY OUTCOMES:
descriptive phenomenological research method | post-test at Week 8
  Each interview should not exceed 90 minutes and should be recorded using recording equipment. Qualitative research methods are quite suitable for exploring or less explored research areas or topics, and can gain insight into the nature, characteristics and attributes of life situations, life events, and life experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan-Yi Huang, DNSc, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Xuan-Yi Huang, Taipei, Peitou, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bry K, Bry M, Hentz E, Karlsson HL, Kyllonen H, Lundkvist M, Wigert H. Communication skills training enhances nurses' ability to respond with empathy to parents' emotions in a neonatal intensive care unit. Acta Paediatr. 2016 Apr;105(4):397-406. doi: 10.1111/apa.13295. Epub 2016 Jan 21. PMID 26648201
- [Background] Cao X, Chen L. The impact of empathy on work engagement in hemodialysis nurses: The mediating role of resilience. Jpn J Nurs Sci. 2020 Jan;17(1):e12284. doi: 10.1111/jjns.12284. Epub 2019 Jul 29. PMID 31359610
- [Background] Derksen F, Bensing J, Lagro-Janssen A. Effectiveness of empathy in general practice: a systematic review. Br J Gen Pract. 2013 Jan;63(606):e76-84. doi: 10.3399/bjgp13X660814. PMID 23336477
- [Background] Fleming BD, Thomas SE, Burnham WS, Charles LT, Shaw D. Improving Ethnocultural Empathy in Healthcare Students through a Targeted Intervention. J Cult Divers. 2015 Summer;22(2):59-63. PMID 26245011
- [Background] Kahriman I, Nural N, Arslan U, Topbas M, Can G, Kasim S. The Effect of Empathy Training on the Empathic Skills of Nurses. Iran Red Crescent Med J. 2016 Jun 5;18(6):e24847. doi: 10.5812/ircmj.24847. eCollection 2016 Jun. PMID 27621922